CLINICAL TRIAL: NCT01708499
Title: Feasibility Study: Evaluation of the Ulthera® System for Efficacious and Safe Treatment of Laxity/Crepiness and Texture of Abdominal Tissue
Brief Title: Feasibility Study: Evaluation of the Ulthera® System for Treatment of Abdominal Tissue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: ULT-128
Record Dates: First submitted 2012-10-15; First posted 2012-10-17 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2013-06

CONDITIONS: Skin Laxity; Skin Crepiness
Keywords: Ulthera® System; Ultherapy™ Treatment; Ulthera, Inc.; Ultrasound treatment for skin tightening
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study treatment (Experimental): All enrolled subjects will receive one Ulthera System Treatment.
  Interventions: Device: Ulthera System Treatment

INTERVENTIONS:
Device: Ulthera System Treatment — Focused ultrasound energy delivered below the surface of the skin
  Other Names: Ultherapy™

SUMMARY:
Enrolled subjects will receive one UltherapyTM treatment on the abdomen. Follow-up visits will occur at 90 and 180 days post-treatment. Study images will be obtained pre-treatment, immediately post-treatment, and at each follow-up visit.

DETAILED DESCRIPTION:
This is a prospective, single-center, pilot clinical trial to evaluate the efficacy of the Ulthera® System for improving laxity/crepiness and texture of abdominal tissue. Changes from baseline in the laxity, crepiness and texture of abdominal skin will be assessed at each study follow-up visit. Global Aesthetic Improvement Scale scores, assessments of dermal thickness, and patient satisfaction questionnaires will also be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 25 to 60 years.
* Subject in good health.
* Skin laxity in the abdomen
* Understands and accepts the obligation not to undergo any other procedures in the areas to be treated through the follow-up period.
* Willingness and ability to comply with protocol requirements, including returning for follow-up visits and abstaining from exclusionary procedures for the duration of the study.

Exclusion Criteria:

* Presence of an active systemic or local skin disease that may affect wound healing.
* Severe solar elastosis.
* Excessive subcutaneous fat in the abdomen.
* Excessive skin laxity on the abdomen.
* Significant scarring in areas to be treated.
* Open wounds or lesions in the area to be treated.
* Inability to understand the protocol or to give informed consent.
* BMI equal to and greater than 30.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-03; Primary Completion 2013-01 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Improvement laxity/crepiness and texture of abdominal tissue | 90 days post-treatment
  Determined by a masked, qualitative assessment of photographs at 90 days post treatment compared to baseline

SECONDARY OUTCOMES:
Overall aesthetic improvement | 180 days post-treatment
  The Global Aesthetic Improvement Scale scores will be obtained from the investigator and subject, comparing post-treatment photos to pre-treatment photos.

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Sasaki, MD, Principal Investigator
Locations (1):
- Sasaki Advanced Aesthetic Medical Center, Pasadena, California, United States